CLINICAL TRIAL: NCT04705051
Title: Multicenter, Open-label, Extension Study to Characterize the Long-term Efficacy and Safety of Early Versus Delayed Treatment With Venglustat (GZ/SAR402671) in Patients at Risk of Rapidly Progressive Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Long-term Treatment of Autosomal Dominant Polycystic Kidney Disease (ADPKD) With Venglustat
Acronym: STAGED-PKD-EXT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: LTS15823 (long-term extension of the EFC15392 study) was stopped after protocol specified interim analysis for futility of the parent EFC15392 study met the prespecified stopping rule based on the primary outcome measure.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS15823; 2020-004400-34 (EudraCT Number); U1111-1256-8805 (Other: UTN)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Congenital Cystic Kidney Disease
MeSH Terms: conditions — Kidney Diseases, Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venglustat (Experimental): Participants were to be treated with venglustat 15 milligrams once daily orally for 24 months or until venglustat was commercially available, whichever came first.
  Interventions: Drug: Venglustat GZ402671

INTERVENTIONS:
Drug: Venglustat GZ402671 — Pharmaceutical form: capsule Route of administration: oral

SUMMARY:
Primary Objective:

-To determine the effect of early versus delayed treatment with venglustat on the total kidney volume (TKV) in participants at risk of rapidly progressive autosomal dominant polycystic kidney disease (ADPKD).

Secondary Objective:

* To determine the effect of early versus delayed treatment with venglustat on the renal function (estimated glomerular filtration rate [eGFR] [Chronic Kidney Disease Epidemiology Collaboration {CKD-EPI} equation]).
* To characterize the safety profile of venglustat.
* To evaluate the effect of venglustat on the lens by ophthalmological examination.
* To evaluate the effect of venglustat on mood using Beck Depression Inventory-II (BDI-II).

DETAILED DESCRIPTION:
The planned study duration per participant was 25.5 months (maximal). Screening period (when applicable): up to 2 weeks. Core treatment period: 24 months. Follow-up: 30 days after final dose of the investigational medicinal product (IMP) (venglustat).

ELIGIBILITY:
Inclusion criteria :

* Male or female adult with ADPKD who had completed the treatment period in Stage 1 or Stage 2 of Study EFC15392 (NCT03523728).
* The participants who had an eGFR >30 mL/min/1.73 m^2:

  1. Measured at Visit 11 of the EFC15392 study for participant enrolled in the LTS15823 study at the time of Visit 12 (Month 24; end-of treatment visit) of the EFC15392 study.
  2. Measured at Screening visit for participant enrolled in the LTS15823 study not concomitantly to the Visit 12 (Month 24; end-of treatment visit) of the EFC15392 study.
* Contraceptive used by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Male participants who agreed to practice true abstinence in line with their preferred and usual lifestyle or to use double-contraceptive methods for the entire duration of the study and for at least 90 days following their last dose of IMP.
  2. Female participants who had a negative urine pregnancy test at the Baseline visit and agreed to practice true abstinence in line with their preferred and usual lifestyle or to use double contraceptive methods (including a highly effective method of contraception) for the entire duration of the study and for at least 6 weeks following their last dose of IMP.
* Capable of giving signed informed consent before performance of any study related procedures not part of standard medical care.
* Able to read, comprehend, and respond to the study questionnaires.

Exclusion criteria:

* For participants who had lag phase between the end of the EFC15392 study and Screening visit (Visit 0) in the LTS15823 study.
* The participant had a new clinically significant, uncontrolled medical condition that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or which would affect the efficacy or safety analysis if the condition exacerbated during the study, or that might significantly interfere with study compliance, including all prescribed evaluations and follow-up activities.
* A history of drug abuse and/or alcohol abuse or alcohol dependence during the lag phase between the end of the EFC15392 study and Screening visit (Visit 0) in the LTS15823 study when applicable.
* Administration of tolvaptan or other polycystic kidney disease-modifying agents (somatostatin analogues) within 3 months prior to the Screening visit (Visit 0) in the LTS15823 study when applicable.
* The participant was currently receiving potentially cataractogenic medications, including a chronic regimen (more frequently than every 2 weeks) of any route of corticosteroids (including medium and high potency topical steroids), or any medication that may cause cataract, according to the Prescribing Information.
* The participant had received strong or moderate inducers or inhibitors of CYP3A4 within 14 days or 5 half lives, whichever was longer, prior to the Baseline visit (including consumption of grapefruit-containing products within 72 hours of starting venglustat administration).
* Participation in another investigational interventional study or use of IMP, within 3 months or 5 half-lives, whichever was longer, before the Baseline visit (Visit 1) except participation in the EFC15392 study when applicable.
* Liver enzymes (alanine aminotransferase /aspartate aminotransferase) or total bilirubin >2 times the upper limit of normal unless the participant had the diagnosis of Gilbert syndrome. Participants with the Gilbert syndrome should had no additional symptoms or signs which suggest hepatobiliary disease and serum total bilirubin level no more than 3 milligrams per decilitre (mg/dL) (51 micromoles per litre [μmol/L]) with conjugated bilirubin less than 20 percent (%) of the total bilirubin fraction.

For participants with or without lag phase between the end of EFC15392 study and entry into LTS15823 study:

* The participant was pregnant or lactating.
* Presence of severe depression as measured by BDI-II >28 at Visit 1 (for participants enrolled in the LTS15823 study at the time of the end of treatment visit of the EFC15392 study) or at Visit 0 (for participants enrolled in the LTS15823 study after the end-of-treatment visit of the EFC15392 study).
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Investigational Site Number :8400019, Morgantown, West Virginia, United States
- Investigational Site Number :0360001, Westmead, New South Wales, Australia
- Investigational Site Number :0560002, Leuven, Belgium
- Investigational Site Number :2760001, Berlin, Germany
- Japan (4):
  - Investigational Site Number :3920001, Sapporo, Hokkaido
  - Investigational Site Number :3920007, Osaka, Osaka
  - Investigational Site Number :3920002, Bunkyo-ku, Tokyo
  - Investigational Site Number :3920004, Shinjuku-ku, Tokyo
- Investigational Site Number :5280002, Nijmegen, Netherlands
- Investigational Site Number :4100002, Seoul, Seoul-teukbyeolsi, South Korea
- Investigational Site Number :7240003, Barcelona, Barcelona [Barcelona], Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS15823 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25299&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 centers in 8 countries. A total of 24 participants were enrolled in the study between 09 February 2021 and 13 July 2021. Out of which, 23 participants were treated.
Pre-assignment Details: Participants at risk of rapidly progressive autosomal dominant polycystic kidney disease (ADPKD) who had previously completed Stage 1 of Study EFC15392 (NCT: NCT03523728) were enrolled in this study.
Groups:
- Venglustat 15mg: Participants received open-label treatment with Venglustat 15 milligrams (mg) once daily orally up to a maximum of 16 weeks.
Period: Overall Study
Arm/Group | Venglustat 15mg
Started | 24
Treated | 23
Completed | 0
Not Completed | 24
Not completed — Enrolled but not treated | 1
Not completed — Study terminated by sponsor | 23

BASELINE CHARACTERISTICS:
Population: Analysis was performed on enrolled population which included all participants allocated to an intervention kit by interactive response technology (IRT) regardless of whether the intervention was received or not.
Groups:
- Venglustat 15mg: Participants enrolled in open-label Venglustat 15 mg once daily orally.
Arm/Group | Venglustat 15mg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Kidney Volume (TKV)
Description: Total kidney volume is a measure of disease progression in the ADPKD participants. Study LTS15823 was terminated prematurely by the Sponsor following a decision to terminate the parent study EFC15392 (NCT03523728). Study EFC15392 was terminated based on the results of the planned prespecified futility analysis performed for this study. Termination decision was due to a lack of efficacy in the ADPKD population and not linked to safety findings with venglustat. Due to the early termination of study LTS15823 and low enrollment numbers, efficacy analysis was not performed.
Time Frame: From the EFC15392 study Baseline to 24 months of open-label extension study LTS15823
Population: For study LTS15823, due to low number of enrollments as compared to the planned numbers and very limited data available post-baseline (only 2 participants reached the planned Month 3 visit), the analysis was carried out only on the available safety and tolerability data. Due to early termination of the study, no efficacy data was available at Month 24 hence the efficacy analysis was not performed.
Arm/Group | Venglustat 15mg
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From the Baseline in Estimated Glomerular Filtration Rate (eGFR) as Assessed by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Description: eGFR is a measure of kidney function assessed through blood/serum. Study LTS15823 was terminated prematurely by the Sponsor following a decision to terminate the parent study EFC15392 (NCT03523728). Study EFC15392 was terminated based on the results of the planned prespecified futility analysis performed for this study. Termination decision was due to a lack of efficacy in the ADPKD population and not linked to safety findings with venglustat. Due to the early termination of study LTS15823 and low enrollment numbers, efficacy analysis was not performed.
Time Frame: From the EFC15392 study Baseline to 24 months of open-label extension study LTS15823
Population: as for outcome 1
Arm/Group | Venglustat 15mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in participant who received investigational medicinal product (IMP) and did not necessarily have a causal relationship with treatment. All reported AEs were TEAEs that developed/worsened during 'TEAE period' (defined as the time from the first administration of the IMP in LTS15823 study up to the last IMP administration + 30 days). A SAEs was defined as any AE that at any dose results in: death; is life threatening; requires initial or prolonged inpatient hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via an authorized medicinal product; is a medically important event.
Time Frame: From the first administration of the IMP in LTS15823 study up to the last IMP administration in LTS15823 study + 30 days (i.e., up to approximately 20 weeks)
Population: Analysis was performed on Long-term extension safety population which included all participants who had received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Venglustat 15mg: Participants received open-label treatment with Venglustat 15 mg once daily orally up to a maximum of 16 weeks.
Arm/Group | Venglustat 15mg
Number analyzed (Participants) | 23
Participants
  Any TEAEs | 2
  SAEs | 1

4. Secondary Outcome: Change From Baseline in Lens Clarity During the Open-label Extension Treatment-emergent Period of LTS15823 Study
Description: Change from EFC15392 study Baseline in the lens clarity was assessed by ophthalmological examination with World Health Organization (WHO) simplified cataract grading system during the open label extension treatment-emergent period of LTS15823 study. Study LTS15823 was terminated prematurely by the Sponsor following a decision to terminate the parent study EFC15392 (NCT03523728). Study EFC15392 was terminated based on the results of the planned prespecified futility analysis performed for this study. Termination decision was due to a lack of efficacy in the ADPKD population and not linked to safety findings with venglustat. Baseline was defined as the values from EFC15392 study Baseline.
Time Frame: Baseline (EFC15392 study Baseline); from first administration of IMP up to last administration of IMP of open-label extension study LTS15823 + 30 days (i.e., up to approximately 20 weeks), in comparison to the EFC15392 study Baseline
Population: For study LTS15823, due to early termination of the study, no ophthalmological data was collected at the planned visits as per protocol and thus the planned analysis was not performed.
Arm/Group | Venglustat 15mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Effect on Mood With Change From Baseline in Beck Depression Inventory (BDI-II) Score During the Open-label Extension Treatment-emergent Period of LTS15823 Study
Description: BDI-II was a validated self-reported instrument of 21 questions which were each scored on a Likert scale of 0 to 3. Total score was calculated as sum of all scores of 21 questions. Total scores ranged from 0 (minimal depression) to 63 (severe depression), with higher score totals indicating more severe depression symptoms (0 to 13: indicates minimal depression;14 to 19: indicates mild depression; 20 to 28: indicates moderate depression; and 29 to 63: indicates severe depression). A negative change from baseline indicated an improvement. Baseline was defined as the values from EFC15392 study Baseline.
Time Frame: Baseline (EFC15392 study Baseline); from first IMP administration up to 3 months in study LTS15823, in comparison to the EFC15392 study Baseline
Population: Analysis was performed on long-term extension safety population. BDI score was collected for 16 participants at Baseline and up to 3 months at the end of trial visit i.e., within 30 days after last dose of study drug following the decision for early termination of the study. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venglustat 15mg
Number analyzed (Participants) | 16
score on a scale
  Baseline | 2.188 (4.086)
  Change from Baseline | -0.875 (4.455)

ADVERSE EVENTS:
Time Frame: From the first administration of the IMP in LTS15823 study up to the last IMP administration in LTS15823 study + 30 days (i.e., up to approximately 20 weeks)
Description: Reported AEs were TEAEs i.e., AEs that developed/worsened during the 'TEAE period'. Analysis was performed on long-term extension safety population.
Arm/Group | Venglustat 15mg
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venglustat 15mg (N=23)
Wound Infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the Sponsor following a decision to terminate the parent study EFC15392. Termination decision was due to lack of efficacy in ADPKD population and not linked to safety findings with venglustat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT04705051/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT04705051/SAP_001.pdf